CLINICAL TRIAL: NCT05998811
Title: Exploring Uterine Cancer Clinical Trials - Revealing Participation Patterns in Individuals With Uterine Cancer
Brief Title: Insights Into Participating in Studies for Uterine Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 82665307
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Uterine Cancer
Keywords: Uterine Cancer
MeSH Terms: conditions — Uterine Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical study participation has historically been heavily biased toward specific demographics.

Several people will be invited to enroll in this trial so that it may collect a variety of data about uterine cancer clinical study experiences and identify barriers to participation as well as the causes of participants' failure or withdrawal.

People with uterine cancer who are invited to take part in medical study will benefit from the analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old and ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Diagnosis of uterine cancer
* No prior treatment for uterine cancer

Exclusion Criteria:

* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Enrolled in another research study
* Inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Uterine cancer patients who are actively considering enrolling in a clinical trial for the said condition, but have not yet completed enrollment and randomization phases.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to enroll in a uterine cancer clinical research | 3 months
Rate of patients who remain in a uterine cancer clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Filippova OT, Leitao MM. The current clinical approach to newly diagnosed uterine cancer. Expert Rev Anticancer Ther. 2020 Jul;20(7):581-590. doi: 10.1080/14737140.2020.1782750. Epub 2020 Jun 22. PMID 32531179
- [Background] Wang Z, Guo E, Yang B, Xiao R, Lu F, You L, Chen G. Trends and age-period-cohort effects on mortality of the three major gynecologic cancers in China from 1990 to 2019: Cervical, ovarian and uterine cancer. Gynecol Oncol. 2021 Nov;163(2):358-363. doi: 10.1016/j.ygyno.2021.08.029. Epub 2021 Sep 8. PMID 34507827
- [Background] Torres D, Myers JA, Eshraghi LW, Riley EC, Soliman PT, Milam MR. Risk factors for the development of uterine cancer in breast cancer survivors: an army of women study. Ann Surg Oncol. 2015;22(6):1974-9. doi: 10.1245/s10434-014-4193-5. Epub 2014 Nov 1. PMID 25361886

DOCUMENTS (1):
  • Informed Consent Form (2023-08-11): https://cdn.clinicaltrials.gov/large-docs/11/NCT05998811/ICF_000.pdf